CLINICAL TRIAL: NCT07256093
Title: The Effectiveness of Acceptance and Commitment Therapy (ACT) on Dysfunctional Attitudes and Difficulties in Emotion Regulation Among University Students in Malaysia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Wei Jun Tan, Mr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/KK/24080672
Record Dates: First submitted 2025-11-19; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Depression; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Intervention Group (Experimental): Participants in the intervention group attended six weekly individual sessions of ACT intervention (1 hour per session) conducted online via the Webex platform.
  Interventions: Other: Acceptance and Commitment Therapy (ACT)
- Waitlist Control Group (No Intervention): Participants in the control group were placed on a waitlist and completed the same outcome measures at three different time points (week 1, week 3, and week 6). After the completion of data collection, they were then divided into two groups and attended two group sessions of ACT (1.5 hours per session), each covering three of the six ACT main components.

INTERVENTIONS:
Other: Acceptance and Commitment Therapy (ACT) — Six sessions of ACT were conducted
  Session 1:
  Introduction. Theme: Broaden your horizon. Values and value-based actions. Identifying what matters the most in your life and acting accordingly.
  Session 2: Theme: Present moment. Mindfully notice your internal and external experiences, notice the movement of your breath. Live in the present moment. To address difficulties in emotion regulation.
  Session 3: Theme: Cognitive defusion. The power of thoughts. Identify your unwanted thoughts and emotions and learn to describe, name, and welcome them. To address dysfunctional attitudes.
  Session 4: Theme: The observer's stance. Learn to view your thoughts and emotions from an observer's stance. To address difficulties in emotion regulation.
  Session 5: Theme: Toward an attitude of acceptance. Let go of your struggle and learn acceptance towards your wakefulness and unwanted thoughts. To address dysfunctional attitudes.
  Session 6: Theme: Summary of the programme. Plans committed action.
  Arms: ACT Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if Acceptance and Commitment Therapy (ACT) can reduce dysfunctional attitudes and difficulties in emotion regulation among university students in Malaysia.The main questions it aims to answer are:

* Will participants who receive ACT show statistically significant reduction in dysfunctional attitudes scores compared to those in the control group?
* Will participants who receive ACT show statistically significant reduction in difficulties in emotion regulation scores compared to those in the control group?
* Will participants who receive ACT show statistically significant reduction in dysfunctional attitudes scores from pre-test to intermediate-test and from pre-test to post-test?
* Will participants who receive ACT show statistically significant reduction in difficulties in emotion regulation scores from pre-test to intermediate test and from pre-test to post-test?

Researchers will compare ACT group to a waitlist control group to see if ACT work to reduce dysfunctional attitudes and difficulties in emotion regulation.

Participants in the ACT group will

* attend six weekly individual sessions of ACT intervention (1 hour per session) conducted online
* complete the outcome measures at three different time points (week 1, week 3, and week 6)

Meanwhile, participants in the waitlist control group

* will not receive any intervention during the data collection period
* will be asked to complete same outcome measures at three different time points (week 1, week 3, and week 6)

ELIGIBILITY:
Inclusion Criteria:

* (a) Malaysian citizens; (b) currently enrolled as a university student; (c) be proficient in both Malay and English languages; (d) aged between 18 and 32 years old; (e) reported mild to moderate depression, anxiety, and/or stress levels according to the DASS-21

Exclusion Criteria:

* (a) reported severe depression, anxiety, and/or stress on the DASS-21; (b) expected to graduate before study ends; (c) had been diagnosed with any psychological disorder prior to the study; (d) were currently receiving psychotherapeutic medication and/or psychological interventions.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation | Baseline, Week 3, and Week 6
  It is measured as the total score on the Difficulties in Emotion Regulation Scale-18 Malay, where a higher score indicates a greater degree of difficulties in emotion regulation.
Dysfunctional Attitudes | Baseline, Week 3, and Week 6
  It is measured as the total score on the Dysfunctional Attitude Scale-Malay, where a higher score indicates a greater degree of dysfunctional attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No